CLINICAL TRIAL: NCT05336084
Title: Center for Adolescent Reward, Rhythms and Sleep Project 1
Brief Title: Circadian Rhythms and Homeostatic Sleep Drive and Their Effect on Reward and Cognitive Control Systems in Adolescents
Acronym: CARRS-P1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Peter Franzen, Associate Professor of Psychiatry and Clinical and Translational Science, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY20030237; P50DA046346 (NIH)
Record Dates: First submitted 2021-08-31; First posted 2022-04-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Sleep
Keywords: adolescence; sleep; substance use; reward sensitivity and motivation; circadian phase and alignment; homeostatic sleep drive; ultradian sleep/wake schedule
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultradian Sleep/Wake protocol (Experimental): This study uses an ultradian sleep/wake protocol to examine circadian and homeostatic sleep systems and their contributions to reward and cognitive control function. All participants will undergo the ultradian sleep/wake protocol following a night of sleep in the lab (measured with polysomnography) for 36 hours. The ultradian sleep/wake protocol will last for 36 h, during which every 120-minutes, there will be an 80-minute period of waking, followed by a 40-minute sleep opportunity. A repeat night of sleep will occur at the end of the 36-hour ultradian sleep/wake protocol.
  Interventions: Behavioral: Ultradian sleep/wake protocol

INTERVENTIONS:
Behavioral: Ultradian sleep/wake protocol — 120-minute schedule, consisting of 80 minutes awake followed by a 40 minute sleep opportunity for 36 hours

SUMMARY:
Adolescence is a time of heightened reward sensitivity and greater impulsivity. On top of this, many teenagers experience chronic sleep deprivation and misalignment of their circadian rhythms due to biological shifts in their sleep/wake patterns paired with early school start times, which may increase the risk for substance use (SU). However, what impact circadian rhythm and sleep disruption either together or independently have on the neuronal circuitry that controls reward and cognition, or if there are interventions that might help to modify these disruptions is unknown. Project 1 (P1), specifically examines homeostatic and circadian characteristics as mechanisms linking habitual sleep patterns, reward and cognitive control (at subjective, behavioral, and circuit levels), and longitudinal substance use risk.

DETAILED DESCRIPTION:
P1 will study 96 adolescents ages 13-15, stratified by habitual sleep timing (early, intermediate, late), in a 60-h laboratory study. Participants will monitor sleep patterns at home for 2 weeks with actigraphy and sleep diary, and will also complete fMRI measures of reward and cognitive control. This will be followed by a 60-hour laboratory visit. The laboratory session includes two nights of polysomnography (PSG) sleep studies, separated by 36 h of an ultradian sleep/wake protocol-every 120-minutes, there will be an 80-minute period of waking, followed by a 40-minute sleep opportunity. Participants will be in dim light conditions and temporal isolation for the first 24 h of the ultradian sleep/wake protocol. Physiological circadian measures include salivary melatonin; core body temperature (CBT); and molecular rhythms from hair follicle cells (examined in Project 3). Physiological sleep homeostatic measures include waking EEG theta power, slow-wave sleep rebound following the 36-h ultradian sleep/wake protocol, and repeated sleep latency on the sleep opportunities. Behavioral tests (Reward Anti-Saccade task to index cognitive control with/without reward modulation; Psychomotor Vigilance Test) and self-reports of mood/sleepiness will be collected every 2 h. Longitudinal on-line surveys will assess substance use every 6 months for the life of the grant.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-15 years
* Currently enrolled in a traditional high-school (not cyber- or home-schooled) [school closures during the COVID-19 pandemic are an exception to this]
* Physically and psychiatrically healthy
* Provision of written informed consent and assent

Exclusion Criteria:

* outside age range above
* have a history of alcohol, cannabis, or illicit drug use in the past month, or greater than monthly use in the past year
* have serious medical or neurological disorders, including history of seizures
* have serious psychiatric disorders (e.g. bipolar disorder and schizophrenia)
* taking antidepressants (SSRIs/SSNIs are OK) or medications known to impact sleep/wake function - some medications may be okay if willing and able to discontinue prior to and/or for laboratory procedures
* have sleep disorders other than insomnia or Delayed Sleep Phase Disorder
* have MRI contraindications (i.e., metal in the body; claustrophobia)
* first degree relative with bipolar disorder
* frequent headaches or migraines
* inability to swallow pills/capsules.
* pregnancy
* participants with observed Obstructive Sleep Apnea via Apnealink, as indicated by an Apnea Hypopnea Index (AHI) of greater than 5
* Less than 80 lbs. or a BMI of greater than 35

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in EEG delta power across overnight polysomnography on the night preceding vs. following the 36-hour ultradian sleep/wake protocol. | The first night of sleep preceding the 36-hour ultradian sleep/wake protocol vs the night of sleep following the ultradian sleep/wake protocol
  Change in the slope of EEG delta power (0.5 - 4 Hz) across NREM periods (frontal leads) on the night preceding vs. following the 36-h ultradian sleep/wake protocol (as measured by polysomnography).
Change in slope of waking EEG theta power | Every 2 hours during the 36-hour ultradian sleep/wake protocol
  Assessed every 2 hours across the 36-hour ultradian sleep/wake protocol
Melatonin onset | The first 24-hours of the ultradian sleep/wake protocol
  Endogenous circadian phase estimate of the rise in evening melatonin levels from saliva samples collected over a 24-hour period (every 30 - 60 minutes) under dim light conditions.

SECONDARY OUTCOMES:
Circadian pattern of Core Body Temperature (CBT) | Measured continuously across the 36-hour ultradian sleep/wake protocol.
  Minimum of CBT
Melatonin amplitude | Collected every 30-60 minutes across the first 24-hours of the ultradian sleep/wake protocol
  Amplitude of the 24-hour melatonin period to estimate endogenous circadian phase
Sleep latency | During the 40-minute sleep opportunities collected every two hours across the 36-hour ultradian sleep/wake protocol.
  Time until sleep onset (first 30-second epoch of N2 sleep) as assessed by polysomnography
Influence of sleep and circadian measures on neural correlates of impulse control | Measures from the 36-hour ultradian sleep/wake protocol in relation to an fMRI scan measured 1 to 2 weeks earlier.
  This outcome will be measured during the Stop Signal Task, which is a computerized an fMRI behavioral task. It will be assessed by activation within the Executive Control Network, specifically, activation is defined as bold signal in regions of the Executive Control Network (particularly the inferior frontal gyrus) on correct Stop trials versus correct Go trials.
Influence of sleep and circadian measures on neural correlates of reward anticipation and reward outcome. | 1 to 2 weeks before to immediately after the 36-hour ultradian sleep/wake protocol.
  This outcome will be measured during the Money Incentive Delay Task, which is a computerized an fMRI behavioral task. It will be assessed by activation within the reward network, specifically, activation is defined as bold signals in regions of the reward network (particularly the ventral striatum) on reward anticipation trials versus no money trials.
Performance on the Psychomotor Vigilance Task | 1 to 2 weeks before to immediately after the 36-hour ultradian sleep/wake protocol.
  This outcome will be measured during the Psychomotor Vigilance Task, specifically lapses (reaction times > 500 ms) on this sustained attention task.
Performance on the Reward Anti-Saccade task | Measures collected every two hours during the 36-hour ultradian sleep/wake protocol.
  This outcome will be measured during the Reward Anti-Saccade task, which measures the ability to look away from a target (an anti-saccade).
Substance use | Every 6 months for the duration of the study, up to 4.5 years
  Frequency-based self-reports of substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Franzen, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Current and future investigators, both internal and external, may have access to de-identified data; however only group data would be shared.